CLINICAL TRIAL: NCT07292155
Title: Investigation of the Prevalence of Type D Personality and Stigma in Patients With Cervical Myofascial Pain Syndrome
Brief Title: Type D Personality, and Stigma in Myofascial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Collaborators: Bozok University (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 2025-GOKAEK-2513_2025.07.02505
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cervical Myofascial Pain Syndrome; Chronic Neck Pain; Type D Personality; Psychological Distress; Stigma; Anxiety and Depression; Quality of Life
Keywords: Myofascial Pain Syndrome; Cervical Pain; Chronic Pain; Type D Personality; Distressed Personality; Negative Affectivity; Social Inhibition; Psychological Factors; Stigma; Anticipated Stigma; Chronic Illness Stigma; Anxiety; Depression; Neck Disability; Health-Related Quality of Life; Pain Psychology; Psychosocial Factors; Biopsychosocial Approach
MeSH Terms: conditions — Social Stigma; Anxiety Disorders; Depression; Myofascial Pain Syndromes; Neck Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical Myofascial Pain Syndrome Group: This group includes adults between 18 and 65 years of age who were clinically diagnosed with cervical myofascial pain syndrome for at least six months. Participants were evaluated at the Departments of Neurology and Physical Medicine and Rehabilitation at Bozok University. Each participant completed a detailed clinical and psychosocial assessment using standardized questionnaires, including the Headache Impact Test, the Neck Disability Index, the Hospital Anxiety and Depression Scale, the Type D Personality Scale, the Chronic Illness Anticipated Stigma Scale, and the Short Form 36 Health Survey. These assessments were used to evaluate pain severity, neck-related disability, emotional status, personality traits, perceived stigma, and quality of life.
- Healthy Control Group: This group includes healthy volunteers who were matched to the patient group by age, sex, and education level. Individuals in this group did not have any musculoskeletal, rheumatologic, neurological, or psychiatric disorders. They completed the same assessment battery as the patient group, including the Headache Impact Test, the Neck Disability Index, the Hospital Anxiety and Depression Scale, the Type D Personality Scale, the Chronic Illness Anticipated Stigma Scale, and the Short Form 36 Health Survey, in order to allow direct comparison of psychological and functional characteristics between groups.

SUMMARY:
Cervical myofascial pain syndrome is a chronic musculoskeletal condition characterized by the presence of sensitive trigger points and taut muscle bands, resulting in localized or referred pain, muscle stiffness, and limited range of motion. The disorder frequently leads to functional limitations and a reduction in quality of life. Although the physical features of cervical myofascial pain syndrome have been well documented, its psychological and social dimensions have not been adequately explored. Personality traits and social factors may influence pain perception, coping mechanisms, and treatment adherence. Type D personality, also known as distressed personality, is defined by the coexistence of negative emotions and social inhibition and has been associated with worse outcomes in various chronic diseases. Stigma represents another psychosocial factor that may contribute to disability and emotional distress in chronic pain conditions.

This case-control study aims to investigate the prevalence of Type D personality traits and anticipated stigma among patients with cervical myofascial pain syndrome compared with healthy individuals. The study further explores the relationships between personality type, stigma, and clinical and psychological parameters, including anxiety, depression, disability, and health-related quality of life. Findings are expected to support a more comprehensive, biopsychosocial understanding of cervical myofascial pain syndrome and emphasize the importance of psychological screening and social support in clinical management.

DETAILED DESCRIPTION:
Cervical myofascial pain syndrome is a non-inflammatory pain disorder associated with painful trigger points in skeletal muscles of the neck and shoulder region. It is characterized by regional pain, restricted neck mobility, muscle tightness, fatigue, and autonomic symptoms such as increased sweating or dizziness. The condition is common among adults, particularly women, and often coexists with other chronic pain syndromes such as tension-type headache or fibromyalgia. Because there are no specific laboratory or imaging tests, diagnosis is based on detailed clinical examination and symptom evaluation. The persistence of pain can lead to emotional distress, sleep disturbance, and significant impairment in daily activities.

Personality and psychosocial factors are known to play important roles in chronic pain perception and coping. Type D personality, defined by the presence of both negative affectivity and social inhibition, has been shown to negatively influence health behaviors and quality of life in several chronic disorders. Individuals with this personality type tend to experience anxiety, irritability, and social withdrawal, which may exacerbate pain-related disability and emotional burden. Another relevant factor is stigma, which refers to social devaluation or exclusion based on illness. Patients with chronic pain may internalize stigma, leading to shame, reduced help-seeking behavior, and decreased treatment adherence. Despite its relevance, stigma has not been investigated in patients with cervical myofascial pain syndrome. This study seeks to fill that gap by assessing both Type D personality and anticipated stigma in this patient population.

Materials and Methods

This case-control study was conducted between July 2025 and October 2025 at the Departments of Neurology and Physical Medicine and Rehabilitation, Bozok University Faculty of Medicine, Yozgat, Turkey. Ethical approval was obtained from the Bozok University Clinical Research Ethics Committee (Approval No: 2025-GOKAEK-2513_2025.07.02_505). All participants provided written informed consent before inclusion.

Participants

The study included outpatients aged 18 to 65 years who were clinically diagnosed with cervical myofascial pain syndrome for at least six months. Diagnosis was made according to established clinical criteria, including localized pain at rest, referred pain from a palpable taut band, a hypersensitive tender spot within the affected muscle, and restricted range of motion. The control group consisted of healthy volunteers matched by age, sex, and education level. Exclusion criteria included systemic diseases, rheumatologic or neurologic disorders, psychiatric conditions such as schizophrenia or bipolar disorder, cervical disc herniation, radiculopathy, myelopathy, and use of psychotropic medication.

Data Collection and Instruments

Demographic and clinical data were recorded using a structured questionnaire that included information on age, sex, marital status, educational level, occupation, and disease duration. Participants completed a set of standardized, validated instruments administered face-to-face by trained healthcare professionals:

Headache Impact Test (HIT-6): Assesses the degree to which headaches affect daily activities, including pain intensity, social and cognitive functioning, and emotional well-being. Higher scores indicate greater impact.

Neck Disability Index (NDI): Measures the extent to which neck pain interferes with everyday activities such as reading, working, sleeping, and recreation.

Hospital Anxiety and Depression Scale (HADS): Evaluates symptoms of anxiety and depression over the previous week through two subscales.

Type D Personality Scale (TDPS): A 14-item instrument assessing negative affectivity and social inhibition. Scores equal to or higher than ten on both subscales indicate the presence of Type D personality traits.

Chronic Illness Anticipated Stigma Scale (CIASS): A 12-item scale assessing expected stigma from family and friends, the workplace, and healthcare providers. Each item is rated on a five-point Likert scale, with higher scores representing greater perceived stigma.

Short Form-36 Health Survey (SF-36): Evaluates health-related quality of life across eight domains, including physical functioning, vitality, social functioning, and mental health. Higher scores denote better perceived health status.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 65 years.

Patients diagnosed with cervical myofascial pain syndrome according to Travell and Simons criteria:

1. localized pain at rest,
2. referred pain or altered sensation in the typical referral zone of a trigger point,
3. a palpable taut band containing a hypersensitive tender spot, and
4. restricted range of motion of the affected muscle.

Duration of symptoms for at least six months.

Outpatients followed in the Department of Physical Medicine and Rehabilitation.

Voluntary participation and provision of written informed consent.

Healthy control participants matched by age, sex, and education, without musculoskeletal or systemic diseases.

Exclusion Criteria:

History of cervical disc herniation, radiculopathy, or myelopathy.

Presence of systemic or rheumatologic diseases.

Current psychiatric or neurological disorders such as schizophrenia, bipolar disorder, dementia, epilepsy, autism, or intellectual disability.

Use of psychotropic medication or ongoing psychiatric treatment.

History of major surgery or trauma involving the cervical region.

Pregnancy or lactation.

Inability to complete questionnaires due to cognitive or language barriers.

Refusal or withdrawal of informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult outpatients aged 18-65 years who were diagnosed with cervical myofascial pain syndrome and healthy volunteers matched by age, sex, and education level. All participants were recruited from the Departments of Neurology and Physical Medicine and Rehabilitation at Bozok University Faculty of Medicine. Written informed consent was obtained from each participant after verbal and written explanations of the study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Type D Personality Scale | At baseline
  The Type D Personality Scale is a 14-item self-report instrument assessing two stable personality traits: negative affectivity and social inhibition. Each item is rated on a five-point scale ranging from 0 (false) to 4 (true). Subscale scores range from 0 to 28. Individuals scoring 10 or higher on both subscales are classified as having Type D personality. A validated Turkish version of the scale is available
Chronic Illness Anticipated Stigma Scale | At baseline
  The Chronic Illness Anticipated Stigma Scale is a 12-item questionnaire measuring anticipated stigma across three domains: family and friends, work environment, and healthcare providers. Each item is rated on a five-point Likert scale ranging from 1 (very unlikely) to 5 (very likely). Subscale scores range from 4 to 20, and total scores range from 12 to 60, with higher scores indicating greater perceived stigma. A validated Turkish version of the scale is available.

SECONDARY OUTCOMES:
Headache Impact Test | At baseline
  The Headache Impact Test consists of six items evaluating the impact of headache on daily functioning, including pain severity, role limitations, social functioning, vitality, cognitive functioning, and psychological distress. Each item is scored from 6 to 13, resulting in a total score ranging from 36 to 78. Higher scores indicate greater headache-related impact. A validated Turkish version of the test is available.
Neck Disability Index | At baseline
  The Neck Disability Index is a 10-item questionnaire assessing the impact of neck pain on activities of daily living such as reading, work, sleep, and recreation. Each item is scored from 0 (no disability) to 5 (complete disability), yielding a total score between 0 and 50. Higher scores indicate greater disability. A validated Turkish version of the index is available.
Hospital Anxiety and Depression Scale | At baseline
  The Hospital Anxiety and Depression Scale is a 14-item questionnaire consisting of two subscales that assess anxiety and depression symptoms. Each item is scored from 0 to 3, producing subscale scores ranging from 0 to 21. Higher scores indicate greater symptom severity. A validated Turkish version of the scale is available.
Short Form 36 Health Survey | At baseline
  The Short Form 36 Health Survey is a generic 36-item instrument that evaluates health-related quality of life across eight domains, including physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Domain scores range from 0 to 100, with higher scores reflecting better perceived health status. A validated Turkish version of the survey is available.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be made available upon reasonable request from qualified researchers. The shared data will include variables used for statistical analyses, demographic information, and scale scores collected during the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and related materials will be available beginning 6 months after publication of the article and will remain accessible for 3 years following publication.
Access Criteria: Researchers who submit a reasonable request describing a methodologically sound proposal for data use may obtain access to de-identified data. Requests should be directed to the corresponding author at the email address listed in the publication. Data will be shared electronically via secure file transfer after approval of the request.
URL: https://hastane.bozok.edu.tr

REFERENCES:
- [Background] Kocyigit, H., Turkish validity and reliability of short-form 36. Drug Treat, 1999. 12: p. 102-106.
- [Background] Tünerir, E., Kronik hastalıklarda beklenen stigma ölçeğinin Türkçe geçerlilik ve güvenilirlik çalışması (Tıpta uzmanlık tezi). Sağlık Bilimleri Üniversitesi, İstanbul, 2019.
- [Background] Öncü, E. and S.K. Vayısoğlu, D Tipi Kişilik Ölçeğinin Türk toplumunda geçerlilik ve güvenirlilik çalışması. Ankara Medical Journal, 2018. 18(4): p. 646-656.
- [Background] Aydemir, O., Hastane anksiyete ve depresyon olcegi Turkce formunun gecerlilik ve guvenilirligi. Turk Psikiyatri Derg., 1997. 8: p. 187-280.
- [Background] Telci EA, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagli N. The cultural adaptation, reliability, and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1732-5. doi: 10.1097/BRS.0b013e3181ac9055. PMID 19770615
- [Background] Dikmen PY, Bozdag M, Gunes M, Kosak S, Tasdelen B, Uluduz D, Ozge A. Reliability and Validity of Turkish Version of Headache Impact Test (HIT-6) in Patients with Migraine. Noro Psikiyatr Ars. 2020 Apr 24;58(4):300-307. doi: 10.29399/npa.24956. eCollection 2021. PMID 34924791